CLINICAL TRIAL: NCT04896372
Title: The ACTyourCHANGE Study Protocol: An ACT Based Inter-vention for Adolescents With Obesity: A Randomized Controlled Trial
Brief Title: The ACTyourCHANGE Study Protocol for Adolescents
Acronym: ACTyourCHANGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03C121
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Psychological Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT intervention (Experimental): The ACT condition (comprehensive of standard care) comprises a three-week in-hospital multidisciplinary rehabilitation program for weight loss and a psychological intervention based on ACT combined with a standard psychological assessment and support to the hospitalization.
  Interventions: Other: ACT comprehensive of standard care
- Standard care (Other): The TAU comprises a three-week in-hospital multidisciplinary rehabilitation program for weight loss and the standard psychological assessment and support to the hospitalization
  Interventions: Other: TAU only

INTERVENTIONS:
Other: ACT comprehensive of standard care — The proposed intervention was designed by the authors of the study. It was developed following the main ACT-based manuals, with adjustments according to the users and the context of the study implementation.
  Specifically, we developed a practical and interactive intervention, which comprises practical activities such as roleplay and writing activities and imaginative activities supported by metaphors. The sessions are based on the use of age-appropriate language to convey the most complex therapeutic processes easily. According to Strosahl and colleagues' model, sessions will respectively target the components of openness, awareness, and engagement.
  Arms: ACT intervention
Other: TAU only — adolescents will be assessed by a staff dietician and placed on an individualized hy-pocaloric balanced Mediterranean diet. They will also follow a nutritional counselling aimed at promoting the adoption of a healthy lifestyle. Moreover, they will attend a physical activity program consisting of five training sessions per week lasting one hour each with trainers; In addition, they will be involved in psychological counselling pro-vided once a week by a clinical psychologist, aimed to address psychological factors related to dysfunctional lifestyle habits.
  Arms: Standard care

SUMMARY:
This Randomized Controlled Trial (RCT) aims to evaluate the effectiveness of a brief Acceptance and Commitment Therapy (ACT)-based-intervention combined with treatment as usual (TAU) compared to TAU only in improving psychological conditions in a sample of adolescents with obesity (body mass index, BMI > 97th centile for age and sex). Fifty consecutive adolescents (12-17 years) of both genders with obesity will be recruited among the patients hospitalized in a clinical center for obesity rehabilitation and randomly allocated into two experimental conditions: ACT + TAU vs TAU only. Both groups will attend a three-week in-hospital multidisciplinary rehabilitation program for weight loss. The ACT + TAU condition comprises a psychological intervention based on ACT combined with a standard psychological assessment and support to the hospitalization. The TAU comprises the standard psychological assessment and support to the hospitalization. At pre- to post-psychological intervention participants will complete the Avoidance and Fusion Questionnaire for Youth, the Psychological Well-Being Scale, the Depression Anxiety Stress Scale, the Difficulties in Emotion Regulation Scale, and the Emotional Eating subscale of the Dutch Eating Behavior Questionnaire. Repeated-measures ANOVAs (2x2) will be conducted. The study will assess the effectiveness of a brief ACT-based intervention for adolescents with obesity.

DETAILED DESCRIPTION:
Obesity in childhood and adolescence is becoming a major public health concern. In this respect, recent estimates pointed out that globally 124 million children and adolescents, aged between 5 and 19 years, were obese. In Europe, the prevalence of overweight and obese children and adolescents aged between 5 to 19 years is reported around 19%, with a higher prevalence in southern European countries.

Obesity in children and adolescents is associated with a higher risk of developing several physical and psychological problems that have an impact on their emotional development [3]. Research has reported associations between childhood and adolescent obesity and some form of psychopathology, as depression, anxiety, and attention-deficit/hyperactivity disorder. Besides, children and adolescents with obesity are more likely to suffer from psychosocial disadvantages as discrimination, social isolation, and bullying because of their weight. Moreover, obesity in childhood and adolescence is associated with poor body image, low self-esteem, and low quality of life and well-being.

This evidence suggests that obesity is a complex disease that may dramatically impair psychological health, representing a risk factor for children and adolescents' future development. This aspect calls for a better understanding of the associated risk factors and requires a multidisciplinary approach - entailing medical, nutritional, physical, and psychological components - aimed to address not only weight loss but also improving psychological conditions and treating obesity-related comorbidities.

The development of dysfunctional eating habits is one of the main factors linked to body weight, and it can be considered a barrier to weight loss [14,15]. Evidence from the literature suggests that unhealthy and dysfunctional eating habits could be related to a failure in emotional regulation strategies, that lead individuals to eat in response to difficult emotions, as in case of emotional eating defined as the tendency to eat in response of negative feelings.

Emotional regulation is defined as the ability to manage emotions, which means to recognize, understand, accept and modulate flexible responses to emotions. High emotion regulation allows individuals to act accordingly with personal goals, even in the presence of difficult emotions, while controlling for impulsive behaviors. On the contrary, when emotional regulation is lacking, emotional eating is undertaken to regulate difficult feelings.

Since emotional eating was related to higher consumption of sweet and fatty food, as an attempt to regulate negative feelings, it was found to be positively associated with weight gain and obesity, both in adult and in younger populations.

A theoretical model for explaining disordered eating suggests that momentary stimuli such as the availability of tasty food in the environment, in combination with a modern sedentary lifestyle, accompanied by difficult emotions, can lead people to move toward behaviors perceived to increase or maintain a hedonic state of pleasure, as eating tasty food immediately. The model also suggests that values clarity and behavioral commitment [to connect healthy eating habits to important life values], awareness [of their automatic thoughts], and distress tolerance [negative internal states] are specific self-regulation skills that can help individuals to deal with difficult emotions and control for their behaviors. Such skills are the main focus of Acceptance and Commitment Therapy.

Acceptance and Commitment Therapy (ACT) is a third-wave CBTs raised in the last twenty years. ACT aims to promote psychological flexibility, defined as the ability to live in the "here and now" current moment consciously while implementing behaviors to live in line with one's own values. This can be seen in opposition to experiential avoidance (or psychological inflexibility) which is the attempt to avoid un-pleasant internal states, such as thoughts, feelings, and bodily sensations. The promotion of psychological flexibility is based on three pillars: openness, awareness, and engagement. Openness refers to the willingness to develop an open and acceptable attitude toward one's personal internal states such as thoughts, emotions, and bodily sensations; Awareness refers to the ability to act intentionally with awareness about personal thought and sensations, without automatically reacting; Engagement refers to engage oneself in committed behaviors related to personal values, that is chosen life directions.

Several ACT-based protocols have been successfully applied to adolescents targeting a broad range of conditions, such as cystic fibrosis, chronic pain, ADHD, and at-risk adolescents. In a pilot study conducted by Hayes, Boyd, and Sewell, thirty adolescents referred to a psychiatric outpatient service were randomly assigned to two conditions: in one, they received an ACT intervention; in the other, participants received a standard intervention for depression. The results showed a significant decrease in depressive symptoms in patients undergoing the ACT intervention. In a study conducted by Kemani and colleagues, an ACT-based intervention was applied to adolescents with chronic pain and their family members. Results showed improved acceptance of chronic pain and psychological flexibility in adolescents, as well as decreased depressive symptoms in their parents. ACT has also been applied to adolescents with a post-traumatic stress disorder [30], proving a reduction of symptoms after a 10-week intervention.

Unfortunately, there are not many studies in the literature concerning the application of an ACT protocol for adolescents with overweight/obesity problems. However, evidence suggests that psychological flexibility is an important key factor of psychological health since it allows people to engage in meaningful challenges, in accordance with person's self-concept and important life domains. To the best of our knowledge only one pilot study published in 2019, evaluating the effectiveness of an ACT-based psychological intervention applied in combination with a 16-week lifestyle behavioral modification program in a sample of obese adolescents, was found. This study showed that the intervention was effective in promoting a reduction in BMI and an overall improvement in physical activity and psychological status of obese adolescents. Furthermore, the intervention was positively evaluated by both the adolescents and their parents who participated in the study.

Given these premises, the present study aims to evaluate the effectiveness of a brief ACT-based- psychological intervention, compared to TAU in improving psychological conditions in a sample of adolescents with obesity attending a multidisciplinary rehabilitation program for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI>97th centile according to age- and sex-specific Italian charts;
* Italian mother tongue
* written and informed consent to participate from both parents and written assent from participants

Exclusion Criteria:

* any physical problems or cognitive impairment that could compromise the participation in the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Psychological Well-Being | Change from baseline baseline psychological well-being to 3 weeks
  The Psychological Well-Being Scales (PWB) will be administered to assess psychological well-being. It is a self-report measure that explores six dimensions: self-acceptance, positive relationships with others, autonomy, environmental control, personal growth, and life purpose. The questionnaire consists of 18 items rated on a 4-point Likert scale ranging from 1 ("completely disagree") to 4 ("completely agree"). scre range from 18 to 72. Higher scores indicate higher well-being. The Italian version, assessed for Italian adolescents, is reported to have good psychometric properties (test-retest correlation coefficients: Self-acceptance: r = .82; Positive relationships: r = .81; Autonomy: r = .21; Environmental control: r = .31; Life purpose: r = .81; Personal growth: r = .78.).

SECONDARY OUTCOMES:
Experiential avoidance and fusion | Change from baseline baseline experiential avoidance and fusion to 3 weeks
  The Avoidance and Fusion Questionnaire for Youth (AFQ-Y) will be administered as a measure of experiential avoidance and fusion in adolescents. It consists of 8 items rated on a 5-point Likert scale ranging from 0 ("not at all true") to 4 ("absolutely true"). Scre ranges from 0 to 32. Higher scores indicate higher avoidance and fusion. The Italian version is reported to have moderate internal consistency [Cronbach's alpha =.69] and a good test-retest reliability (r=.64).
Psychological distress. | Change from baseline psychological distress to 3 weeks
  The Depression Anxiety Stress Scale (DASS-21) will be administered as a measure of psychological distress, widely used in samples of adolescents It is a self-report instrument that measures several negative internal states: depression, anxiety, and stress. It consists of 21 items rated on a 4-point Likert scale, ranging from 0 to 3. Scores range from 0 to 63. Higher scores indicate higher distress.The Italian version showed good psychometric properties (Cronbach's Alpha values of subscales ranged from .83 to .91. The Cronbach's Alpha of the total score was = .92).
Emotional regulation | Change from baseline baseline emotional regulation to 3 weeks
  The Difficulties in Emotion Regulation Scale (DERS) will be administered to assess difficulties in emotional regulation. This is a self-report questionnaire consisting of 36 items, rated on a 5-point Likert scale ranging from 1 ("almost never")] to5 ("almost al-ways"). Scores range from 1 to 180. Higher scores indicate greater difficultis in emotional regulation. The Italian version [43], widely used in samples of adolescents is reported to have good psychometric properties (Cronbach's alpha values ranged from .77 to .89. The Cronbach's Alpha of the total score was .92).
Emotional eating | Change from baseline baseline emotional eating to 3 weeks
  The Emotional Eating subscale of the Dutch Eating Behavior Questionnaire (DEBQ) will be administered to assess emotional eating. The DEBQ is a self-report questionnaire used to detect eating behaviors. The Emotional Eating subscale consists of 13 items, rated on a 5-step Likert scale ranging from 0 ("never") to 4 ("almost always"). Scores range from 0 to 52. Higher scores indicate higher emotional eating. The Italian version showed good psychometric properties (Cronbach's Alpha = .97). The DEBQ was chosen as a measure of emotional eating in our sample, since no other validated instruments are available, except for the DEBQ version for parents , unfortunately unsuitable for parents of our sample of hospitalized adolescents

CONTACTS AND LOCATIONS:
Locations (1):
- San Giuseppe Hospital, Istituto Auxologico Italiano IRCSS, Verbania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897
- [Background] Sagar R, Gupta T. Psychological Aspects of Obesity in Children and Adolescents. Indian J Pediatr. 2018 Jul;85(7):554-559. doi: 10.1007/s12098-017-2539-2. Epub 2017 Nov 18. PMID 29150753
- [Background] Giusti EM, Spatola CA, Brunani A, Kumbhare D, Oral A, Ilieva E, Kiekens C, Pietrabissa G, Manzoni GM, Imamura M, Castelnuovo G, Capodaglio P. ISPRM/ESPRM guidelines on Physical and Rehabilitation Medicine professional practice for adults with obesity and related comorbidities. Eur J Phys Rehabil Med. 2020 Aug;56(4):496-507. doi: 10.23736/S1973-9087.20.06232-2. Epub 2020 Apr 15. PMID 32293813
- [Background] Sainsbury K, Evans EH, Pedersen S, Marques MM, Teixeira PJ, Lahteenmaki L, Stubbs RJ, Heitmann BL, Sniehotta FF. Attribution of weight regain to emotional reasons amongst European adults with overweight and obesity who regained weight following a weight loss attempt. Eat Weight Disord. 2019 Apr;24(2):351-361. doi: 10.1007/s40519-018-0487-0. Epub 2018 Feb 16. PMID 29453590
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724